CLINICAL TRIAL: NCT04817579
Title: Dental Photography and Numeric Shade Quantification as a Substitute to Conventional and Instrumental Shade Matching Techniques in the Esthetic Zone: A Controlled Clinical Trial
Brief Title: Dental Photography and Numeric Shade Quantification as a Substitute to Conventional and Instrumental Shade Matching Techniques in the Esthetic Zone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Ahmed Farid Zaki Shehab, Assistant lecturer, Fixed Prosthodontics Department, Cairo University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 39920
Record Dates: First submitted 2021-03-13; First posted 2021-03-26 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Discoloration, Tooth; Chip Tooth; Non Vital Teeth; Trauma Dental
MeSH Terms: conditions — Tooth Discoloration; Tooth Fractures

STUDY DESIGN:
Intervention Model Description: Each patient will try in three crowns with different methods for shade matching.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional visual shade matching (Active Comparator): Patients requiring single crown in the esthetic zone treated with Conventional visual shade matching (Ivoclar Classic shade guide)
  Interventions: Device: Conventional visual shade matching
- Spectrophotometer (Experimental): Patients requiring single crown in the esthetic zone treated with Spectrophotometer (Vita Easy Shade)
  Interventions: Device: Spectrophotometer
- Digital photography combined with eLABor_aid shade analyzing software. (Experimental): Patients requiring single crown in the esthetic zone treated with Digital photography combined with eLABor_aid shade analyzing software.
  Interventions: Device: Digital photography combined with eLABor_aid shade analyzing software

INTERVENTIONS:
Device: Digital photography combined with eLABor_aid shade analyzing software — ELABor_aid is a new approach to objective shade communication and shade reproduction in dentistry, based on numeric quantification obtained from standardized RGB (red-green-blue) images, and the formulation of a patient personal shade recipe using trichromatic subtractive color mixing laws, thus abandoning the use of visual assessment and shade guides entirely. This approach is currently enjoying increasing popularity for its ease of use, reliability as well as for its practically oriented features like its imaging ability or the digital try-in.
  Other Names: eLAB protocol
  Arms: Digital photography combined with eLABor_aid shade analyzing software.
Device: Spectrophotometer — Spectrophotometric measurement methods employing computer calculations, based on color science and theories, allow quantitative evaluation which is objective and appears to be more accurate.
  Other Names: Vita Easy-shade
  Arms: Spectrophotometer
Device: Conventional visual shade matching — Visual shade matching is the most common method, in which a color standard from a commercially available dental shade guide is compared to and matched with the target tooth.
  Other Names: Ivoclar classic shade guide
  Arms: Conventional visual shade matching

SUMMARY:
Visual shade matching is the most common method, in which a color standard from a commercially available dental shade guide is compared to and matched with the target tooth. However, several factors can contribute to perception errors including: different lighting variables, multiple shade systems available in the market with lack of standardization in color systems and corresponding porcelain systems, individual human variables in color perception and lack of understanding of color science.

Therefore, in order to eliminate the uncontrolled variables during the color matching process, instrumental methods have been developed. Spectrophotometric measurement methods employing computer calculations, based on color science and theories, allow quantitative evaluation which is objective and appears to be more accurate. However, extremely high costs, relatively low performance with respect to agreements of the computer-aided devices, and edge loss error make it less acceptable.

One of the most powerful tools in communicating with both patients and dental ceramists is digital photography. Hence, this study is designed to explore the possibilities of a novel approach to shade management (eLABor_aid) utilizing a photocolorimetric (PCM) method and subsequent shade formulation without the use of stock shade guides in comparison to well-known visual and instrumental methods.

The aim of the study is to evaluate the accuracy of digital photography combined with shade analyzing software (eLAB) in optimizing shade matching when compared to conventional and instrumental methods of shade selection.

A Null Hypothesis is suggested where no significant difference regarding shade selection between eLAB protocol, conventional and instrumental methods will be found.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of the patients from 20-50 years old; able to read and sign the informed consent document.
2. Patients able physically and psychologically to tolerate conventional restorative procedures.
3. Patients with no active periodontal or pulpal diseases, having teeth with good restorations.
4. Patients with teeth problems indicated for full coverage restoration (e.g. moderate discoloration, coronal fracture where partial coverage would lack retention, mal-posed or malformed teeth, esthetics enhancement of previously placed crown) where the contralateral/adjacent tooth is present.
5. Patients with root canal treated teeth requiring full coverage restorations even if they need fiber post and core fabrication first.

Exclusion criteria are:

1. Patients with poor oral hygiene and motivation.
2. Patients with teeth with increased incisal translucency.
3. Patients with severe discolored teeth.
4. Patients with smoking habits.
5. Patients with excessive consumption of coffee or tea.
6. Pregnant women to avoid any complication that may occur in dental office due to pregnancy or due to injected anesthetic solution.
7. Patients with psychiatric problems or unrealistic expectation (patient that has phobia from dental treatments or needle injection).
8. Patients suffer from para-functional habits.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Color difference (Delta E) calculated using calibrated images on photoshop software | Immediately after crowns try-in. The crown with the best result will be instantly cemented.
  Photoshop combined with dental photography using Delta E formula. Standardized images will be taken using a standardized protocol and a grey card to calibrate the produced images to ensure standard exposure in all photos. Delta E will be calculated using photoshop software.
  Delta E (ΔE) = [(L1 - L2)² + (a1 - a2)² + (b1 - b2)²]1/2

SECONDARY OUTCOMES:
Shade match using modified USPHS criteria | Immediately after Try-in stage. Each crown will be seated in the patient's mouth and a score will be given by a blinded assessor. The crown with the best shade match will be finally cemented.
  Alpha (Excellent): ideal. Bravo (Acceptable): less than ideal but no modifications required Charlie (Acceptable but modifications needed): staining or other shade modifications required.
  Delta (Unacceptable): remake.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt